CLINICAL TRIAL: NCT03162484
Title: Effect of a Physical Activity Group Programme on the Health of People With Chronic Acquired Brain Injury
Brief Title: Physical Activity and Chronic Acquired Brain Injury
Acronym: PASBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Marta Pérez Rodriguez, Principal investigator, Universidad Politecnica de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Universidad Politécnica
Record Dates: First submitted 2016-10-28; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Brain Injuries; Motor Activity; Quality of Life
MeSH Terms: conditions — Brain Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity intervention group (Experimental): The intervention consisted in doing physical activities two to four times per week, each session last 60 minutes. The program includes different activities: swimming, paddle tennis, football and aerobic exercises into the swimming-pool.
  Each session starts with a warm up. The main part of the session is divided into two sections. The first section includes different exercises to improve balance, mobility and coordination. The second section is comprised of communicative and cooperative games. The session finishes with a cool-down.
  Interventions: Behavioral: Experimental group
- Control group (No Intervention): People in control group did not receive any physical activity program.

INTERVENTIONS:
Behavioral: Experimental group — The program includes different activities: swimming, paddle tennis, football and aerobic exercises into the swimming-pool.
  Arms: Physical activity intervention group

SUMMARY:
Most individuals who have survived an acquired brain injury (ABI) present consequences affecting the sensorimotor, cognitive, affective or behavioural components. The conditions can vary from mild to extreme. The consequences of an ABI may have a considerable impact on their functioning, and secondary conditions like depression or sedentary behaviours, so they suffer changes in their Health-Related Quality of Life (HRQoL).

The purpose of this project is to determine the effect of a physical activity group program on HRQoL. As well as to identify factors that facilitate or act as a barrier to practice physical activity.

DETAILED DESCRIPTION:
This study is a quasi experimental pre-post test with nonequivalent group design. There were two groups: 30 subjects with chronic ABI took part in a physical activity group program designed by a Sport Club in Madrid, Spain; and 30 subjects with chronic ABI which did not practice physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with mild to moderate chronic acquired brain injury from any cause.
* Being over 18 years of age.
* Being practice two or more sessions per week.
* Ability to understand and complete questionnaires in Spanish.
* Voluntary participation in the study.
* Signed informed consent by the patient and/or their primary caregiver.

Exclusion Criteria:

* Return to work
* Aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Mood change measurement | Change from baseline mood at 18 weeks
  Profile of Mood States (POMS) Questionnaire
Quality of life change measurement | Change from baseline quality of life at 18 weeks
  Short Form 36 Health Survey
Participation in Physical Activities change measurement | Change from baseline participation at 18 weeks
  Global Physical Activity Questionnaire

SECONDARY OUTCOMES:
Depression change measurement | Change from baseline depression at 18 weeks
  Beck Depression Inventory
Months since injury | Baseline
  sociodemographic data questionnaire
Amount of weekly physical activity | Baseline
  sociodemographic data questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pérez, PhD, Study Director — Universidad Politecnica de Madrid

IPD SHARING:
Plan to Share IPD: Undecided